CLINICAL TRIAL: NCT01407484
Title: Diagnosis and Treatment of Male Infertility Related to Inflammatory Syndrome: Therapeutic Trial
Brief Title: Male Infertility Related With Post Infection Inflammatory Syndrome
Acronym: SIGMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P081215
Record Dates: First submitted 2011-06-30; First posted 2011-08-02 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Male Infertility; Leukopenia; Postinfection Inflammation; Oxidative Stress
Keywords: Infertility; Assisted reproductive technology; Double blind therapeutical trial; Multicentric study; Prospective randomized study
MeSH Terms: conditions — Infertility, Male; Leukopenia; Infertility | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Cortancyl (prednisone) 0,2 mg/kg/day for 3 weeks and 0,1mg/kg/day for 1 week
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — 0,2 mg/kg/day for 3 weeks and 0,1mg/kg/day for 1 week.
  Arms: Treatment
Drug: Placebo — Placebo 0,2 mg/kg/day for 3 weeks and 0,1mg/kg/day for 1 week
  Arms: Placebo

SUMMARY:
BACKGROUND: One couple out of 6 consults for infertility during their sexual life. In 60% of cases a male factor is associated or is the main infertility factor. Inflammatory Syndrome (IS), characterized by the presence of a leukocytospermia is found in 12% of the cases. Leukocyte degranulation causes oxidative stress (OS) through the formation of free radicals attacking the sperm cell functions.

HYPOTHESIS: To establish the responsibility of the IS, and OS, in chronicle inflammatory male infertility, the investigators hypothesize that its treatment (as well as its possible cause) must restore or improve the fertilizing capacity of patients sperm.

METHODS: This prospective randomized study will test the response to the treatment. The investigators shall measure cellular degradation products due to the OS, thereby certifying that it does have a deleterious effect on sperm cell. Seminal biochemistry will also assess the impact of the syndrome on the genital tract glands and follow its evolution.

The patients will be included in the study as soon as the leukocytospermia will be > 0,5*106/ml or as soon as the elastase will be > 500 ng/mL.

The examinations will be performed using flow cytometry, CASA (Computer Assisted Semen Analysis). The analysis of sperm morphology will be centralized.

Primary endpoint will be a reduction in the percentage of 8OH-dG below 35 %. We anticipate that it should arrive to 20 % of the patients included in the arm treatment by corticosteroid therapy. All in all will thus be needed 50 patients in the group placebo and 50 in the group treated.

Secondary endpoint the improvement of the spermatic parameters and the reduction of the fragmentation of the DNA of sperm cells to the treated subjects.

All these biological markers will be evaluated 6 month after the treatment:

* Fragmentation of the spermatic DNA below 37 % during the follow-up in 6 months
* Leukocytospermia and elastase
* Seminal biochemistry
* Other markers of the inflammatory syndrome and oxidative stress (protein carbonyl, 8OHd-Guanosine)
* Possibly the radiological examinations (Ultrasound and MRI of the genital tract)

In addition it would allow us to propose a policy of prevention towards acquired post-infectious male infertility.

DETAILED DESCRIPTION:
Progress of research. Timeframe Search

* Duration of inclusions: 30 months
* Duration of patient follow-up: 7 months
* Total duration of the study: 37 months Within the framework of their coverage in AMP, the barren couples have a consultation with the doctors of the reproduction and one with the biologists. Between these two visits, a spermatic balance assessment (EXAMINATION N°0) is made including a semen culture, a spermogram or a test of migration survival (TMS) and an elastase.

On the occasion of this examination, aliquots for the measure of 8OH-dG, fragmentation of the spermatic DNA and seminal biochemistry will systematically be taken.

Within the framework of this standard balance assessment of infertility, it is possible that an echography and a MRI of the genital ways are prescribed; if it is the case, the data of these examinations will be collected in the case report form. But these examinations will not be specifically asked for the search.

If a leukocytospermia ≥ 0,5*106/ml is discovered or an increase of the elastase ≥ 500 ng / ml, the dosages of 8OH-dG, the fragmentation and the seminal biochemistry will be made.

The patients will then be seen in consultation of biology (CONSULTATION OF BIOLOGY N°0 = visit of inclusion and randomization).

* If the patients present 8OH-dG > 35 %, and that their semen culture is negative, it will be suggested to them being included in the protocol and the randomization will be made that very day; the patients will receive or an anti-inflammatory treatment (Prednisone) is a treatment placebo.
* If 8OH-dG < 35 % it will be suggested to them participating in the study of the follow-up of the spontaneous evolution of the SO and of SI over 6 months.

A first complete balance assessment will be made in 1 month (EXAMINATION N°1) after the beginning of the treatment in the study (Prednisone or placebo) so as to estimate the evolution at the end of the treatment of the inflammatory and oxidative parameters This balance assessment will not be realized at the inclusive but not randomized patient's.

Patients randomized in the study will have laboratory tests including:

* A semen analysis (leukocytospermia)
* A measure of oxidative stress (8OHd guanosine assay - assay of protein carbonyl - DNA fragmentation)
* A seminal biochemistry (acid 1-4)alpha phosphatase, citrate, zinc, fructose, carnitine and glucosidase

A second balance assessment will be asked 6 months (EXAMINATION N°2) after the beginning of the treatment for two reasons: the first reason is that the improvement of the spermatic parameters is slowly made. If a spermatic change settled down during years she is not going to disappear in the fortnight. It is effectively the experience which we have of it.

Besides the spermatogenesis continuing over three months, a new cycle of production of sperm cells can be estimated only more than three months after the treatment. The second reason is that the second offenses of the chronic inflammations of the reproductive organ are extremely frequent and it is to estimate this rate of second offense that the balance assessment will be remotely asked for more by the treatment or in 6 months.

This review will include all tests of initial assessment:

* A semen analysis (leukocytospermia)
* A measure of oxidative stress (8OHd guanosine assay - assay of protein carbonyl - DNA fragmentation)
* A seminal biochemistry (acid 1-4)alpha phosphatase, citrate, zinc, fructose, carnitine and glucosidase
* An ultrasound of the genital tract and genital tract RMI without injection of any compound

This visit will be scheduled for all patients, whether randomized or not. During this visit, the results of tests carried out at 1 month and 6 months after initiation of treatment will be analyzed. The investigator will collect adverse events that occurred since the randomization visit.

Patients who during the examination in 6 months have a very significant improvement in their semen parameters will propose cryopreserving their sperm.

Assays and analysis on the semen Collections of semen will be done in the Laboratory of Reproductive Biology of each participating centre of research.

Most assays and analysis will be centralized at the Cochin Hospital. Measurement of elastase Elastase assays will be centralized in the Laboratory of Reproductive Biology, Hospital Cochin. The assays will be carried out from 150 µl total sperm collected after liquefaction and frozen at -20 ° C.

Migration Survival Test (MST) This test will be done locally in each participating centre. A smear slide will be made for a centralized analysis of the morphology, to avoid any "centre" effects.

Seminal Biochemistry The biochemical seminal will be centralized in the Laboratory of Biochemistry, Hospital Cochin. This assay, carried out on total sperm collected after liquefaction, including assays of acid phosphatase, citrate, zinc, fructose, carnitine and 1-4.alpha Glucosidase The semen will be collected, centrifuged at 600g for 5 minutes. After centrifugation, 500μl of the supernatant will be frozen at - 20 ° C and used for biochemical seminal.

Measurement of oxidative stress The extent of oxidative stress will be centrally assessed in Cochin Hospital. This assay, carried out on total sperm collected after liquefaction, including the determination of 8OHd-Guanosine, the dosage of protein carbonyl and DNA fragmentation.

The semen will be collected centrifuged at 600g for 5 minutes. After centrifugation:

* 250μl of the supernatant be frozen at - 20 ° C and used for determination of protein carbonyl.
* The pellet will be used for the assay of 8OHdguanosine and DNA fragmentation. Measurement of sperm motion parameters by CASA The measurement of sperm motion parameters by CASA will be performed locally in each participating centre.

Ultrasound and MRI of the genital tract Ultrasounds and MRI will be performed in the genital tract in the central radiology department of hospital Necker.

Conservation of the remaining sample of semen For patients with very significant improvement in their semen parameters during the examination at 6 months, it will be offered self-preservation of semen for any subsequent attempt of ART after the end of the study.

On the other hand, the remaining sample of semen, except if opposition from the patient, will be kept after the end of the research for later use in future research on fertility and inflammation. This collection will be kept at CECOS - Cochin Hospital, Bldg. Cassini - 27 rue du FAUBOURG St Jacques, 75014 Paris under the supervision of Professor Jean-PHILIPPE Wolf.

Stopping rules Patients may discontinue their participation in research if they wish, at any time and for whatever reason, or upon the decision of the investigator. However, the treatment should not be stopped suddenly.

Stopping rules for the participation of a person seeking

* Poor adherence to protocol
* intercurrent disease between the inclusion visit and the visit at 1 month requiring cessation of study. Following the study is that of surveillance.

Procedures for monitoring output test All output tests should be documented and the investigator must specify the reason. For patients considered lost of sight, case report forms should be filled to the last visit. The investigator will make every effort to contact the patient and to know the reason for leaving the trial and his health.

Consequences Patients who quit from the trial will not be re-included in the study. Their numbers are not effectively reused. These patients will still be followed in the non-randomized part of the study.

ELIGIBILITY:
Inclusion criteria :

* Man over 18 years old
* Patient presenting a leukocytospermia ≥ 0,5*106 /ml or an elastase ≥ 500ng/ml
* No infection
* Signed informed consent

Exclusion criteria :

* Patient having less of 106 /ml of sperm cells in the ejaculate
* Patients with diabetes or receiving treatment for diabetes
* Patients already taking anti-inflammatory drugs
* Patients with ongoing anticoagulant therapy
* Patients with history of allergy to anti-inflammatory drug
* Patients with a history of peptic ulcers
* Patient with history of cardiovascular disease (hypertension, cardiac arrhythmia, ...)
* Patients with psychological disorders
* Patient with an infectious condition except for specified indications of Prednisone
* Patients with some evolutional viruses(including hepatitis, herpes, chickenpox, shingles)
* Patient is in a psychotic state still not controlled by treatment
* Patient receiving a live vaccine
* Patients with hypersensitivity to any component of Prednisone
* Patient not affiliated with a social security system

Criteria for randomization

- Patient meeting all inclusion criteria and none of exclusion, and having a 8OH desoxy Guanosine increased ≥ 35%.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-03-02 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2015-05-14 (Actual)

PRIMARY OUTCOMES:
The number of live motile spermatozoa six month after the treatment | 6 months
  Reduction of the percentage of the spermatic 8OH-dG under 35 % to 20 % of the patients between the visit of inclusion / randomization and the visit of follow-up in 6 months

SECONDARY OUTCOMES:
biological markers | 6 months
  Several biological markers will be evaluated 6 months after the treatment, as markers of inflammation and oxidative stress (sperm DNA fragmentation, protein carbonyl, 8OHdGuanosine, leukocytospermia and elastase, seminal biochemistry,ultrasound, and MRI of the genital tract

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Wolf, MD, Phd, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Hospital, Paris, France